CLINICAL TRIAL: NCT04120506
Title: Long Term Impact of Rapid Intravenous Infusion of Velaglucerase Alfa (VPRIV) in Adult Patients With Type 1 Gaucher Disease, Previously on a Stable Dose of VPRIV for at Least 3 Months: an Extension of the Investigator-initiated Study
Brief Title: Long Term Impact of Rapid Intravenous Infusion of Velaglucerase Alfa (VPRIV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Ari Zimran, Professor, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0075-15-SZMC
Record Dates: First submitted 2018-08-10; First posted 2019-10-09 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Gaucher Disease, Type 1
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Intervention Model Description: Objective: To show non-inferiority of rapid (defined as 10') intravenous (IV) infusion versus standard IV infusion rate (60') of VPRIV with regard to safety, pharmacokinetic(PK) profile, and efficacy in patients who have been receiving VPRIV for a minimum of 3 months at a constant dosage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rapid infusion of Vpriv (Experimental): : Infusions at Baseline and during step-wise rate increases and End-of-study will be performed in the Shaare Zedek Medical Center (SZMC) by the Study Nurse who will monitor vital signs (see below) for a total of 8 visits at SZMC. Home therapy will be approved if the patient so desires for 5 infusions in Phase 1 and for the first 5 infusions in Phase 3. All routine hematological and biochemical tests will be performed in the SZMC clinical labs. Abdominal quantitative MR Imaging (MRI) for spleen and liver volumes will be performed at SZMC
  Interventions: Drug: VPRIV

INTERVENTIONS:
Drug: VPRIV — Safety, pharmacokinetics, and efficacy of rapid intravenous infusion of velaglucerase alfa (VPRIV) in adult patients with type 1 Gaucher disease
  Other Names: Velaglucerase Alfa

SUMMARY:
Background: In order to allow our satisfied patients, who have successfully completed 24 months of rapid intravenous infusion of Velaglucerase alfa (VPRIV), to continue with the 10 minutes IV therapy, the clinical trial framework must be extended; and this extension is important for the assessment of long term benefit (up to 5 years) of this regimen of administration of Velaglucerase alfa..

Suggested trial: An additional 36 months home therapy follow up of safety and efficacy of rapid intravenous infusion of Velaglucerase alfa (VPRIV) in adult patients with type 1 Gaucher disease.

Patients must have completed the prior 4 parts / 24 months of the protocol before enrolling into this extension phase ("Part 5") and have provided a new consent before entering PART 5 of the study.

Patients must not have experienced clinically significant AEs, including allergic reactions, in any of the prior study parts of this protocol to be eligible to participate, and have maintained stability in the key disease features.

All infusions of 10' will be given in the context of home therapy. "Clinically significant" AEs will be determined by the PI using standard description of AEs as previously described at phase 3, and if necessary will support withdrawal of the patient from the study.

DETAILED DESCRIPTION:
Every 6 months, patients will be required to come for routine checkups at SZMC, where the following tests will be performed:

* Complete Blood Count (CBC)
* Routine serum biochemistry including liver function tests (LFTs)
* Plasma biomarker lyso Gb-1
* Height & weight & calculation of BMI
* Physical examination and medical history elicited including concomitant medications
* Ultrasound for spleen and liver volumes

In addition, the following tests will be performed at 12, 24 and 36 months:

* Echocardiography
* Electrocardiogram (ECG)
* Urinalysis
* HRQoL questionnaire (TBD)

At each home visit, the following assessments will be performed by the study nurse:

Queries regarding AEs and changes in clinically relevant Gaucher parameters as described by the patient (e.g., bone pain), inter-current illnesses, etc.

Patients will be required to complete the End-of-study visit, including the final infusion at 10', at SZMC. This final visit will include in addition to the usual safety and efficacy assessments and routine tests, (mentioned above) also, DEXA and anti-drug antibodies.

In addition, we would perform a 4th PK measurement at end of the extension period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, non-splenectomized Enzymatic diagnosis & molecular analysis indicative of type 1 Gaucher disease Receiving VPRIV for at least 6 infusions (3 months) prior to Baseline at a constant dose and frequency and without clinically significant AEs including allergic reactions

Exclusion Criteria:

* Experience of a clinically significant AE to VPRIV at any time in the past Existence of a clinically significant co-morbidity

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of change from baseline in blood pressure for rapid infusion-1 | 9 months
  measured by blood pressure pre and post infusion
Incidence of change from baseline in heart rate for rapid infusion-1 | 9 months
  measured by heart rate pre and post infusion
Incidence of change from baseline in temperature for rapid infusion-1 | 9 months
  measured by temperature pre and post infusion

SECONDARY OUTCOMES:
Non deterioration in Gaucher manifestations- stability in platelet counts | 9 months
  Efficacy secondary endpoints are non-deterioration (defined as stability) in platelet count
Non deterioration in Gaucher manifestations- stability in hemaglobin count | 9 months
  Efficacy secondary endpoints are non-deterioration (defined as stability) in hemaglobin count
Non deterioration in Gaucher manifestations- measured by liver volume | 9 months
  Efficacy secondary endpoints are non-deterioration (defined as stability) in organ volumes of liver volume (as previously defined in the TKT034 clinical trial)
Non deterioration in Gaucher manifestations- measured by spleen volumes | 9 months
  Efficacy secondary endpoints are non-deterioration (defined as stability) in organ volumes of spleen volume (as previously defined in the TKT034 clinical trial)
Non deterioration in Gaucher manifestations- measured by lack of elevated biomarker- Lyso-GB1 | 9 months
  Efficacy secondary endpoints are non-deterioration (defined as stability) by lack of sustained increases in the biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Zimran, Principal Investigator — Ari Zimran - Shaare Zedek

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zimran A, Revel-Vilk S, Becker-Cohen M, Chicco G, Arbel N, Rolfs A, Szer J. Rapid intravenous infusion of velaglucerase-alfa in adults with type 1 Gaucher disease. Am J Hematol. 2018 Sep;93(9):E246-E248. doi: 10.1002/ajh.25205. Epub 2018 Aug 9. No abstract available. PMID 29989200